CLINICAL TRIAL: NCT01458275
Title: A 2-Week Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Safety and Efficacy Study of Ciclesonide Nasal Aerosol in Subjects 6 to 11 Years With Seasonal Allergic Rhinitis
Brief Title: A Safety and Efficacy Study of Ciclesonide Nasal Aerosol in Subjects 6-11 Years With Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP060-305
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal Allergic Rhinitis; Ciclesonide; Ciclesonide Nasal Aerosol
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ciclesonide nasal aerosol 37mcg (Active Comparator): ciclesonide nasal aerosol 37mcg - the dose is administered as 1 actuation per nostril to give a total dose of 37 mcg
  Interventions: Drug: Ciclesonide nasal aerosol 37 mcg
- ciclesonide nasal aerosol 74 mcg (Active Comparator): ciclesonide nasal aerosol 74 mcg - the dose is administered as 1 actuation per nostril to give a total dose of 74 mcg
  Interventions: Drug: ciclesonide nasal aerosol 74 mcg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide nasal aerosol 37 mcg — ciclesonide nasal aerosol 37mcg - the dose is administered as 1 actuation per nostril to give a total dose of 37 mcg
  Arms: ciclesonide nasal aerosol 37mcg
Drug: ciclesonide nasal aerosol 74 mcg — ciclesonide nasal aerosol 74 mcg - the dose is administered as 1 actuation per nostril to give a total dose of 74 mcg
  Arms: ciclesonide nasal aerosol 74 mcg
Drug: Placebo — Placebo - one actuation per nostril
  Arms: Placebo

SUMMARY:
This is a 2-week, multicenter, randomized, double-blind, placebo-controlled, parallel group, efficacy and safety study of ciclesonide nasal aerosol administered once daily to male and premenarchal female subjects 6 to 11 years-old diagnosed with SAR.

DETAILED DESCRIPTION:
This is a 2-week, multicenter, randomized, double-blind, placebo-controlled, parallel group, efficacy and safety study of ciclesonide nasal aerosol administered once daily to male and premenarchal female subjects 6 to 11 years-old diagnosed with SAR.

This study will consist of the following:

Screening, Single-blind Placebo Run-in period, Double-blind Treatment period (during this period, subjects will be randomized to double-blind treatment with either ciclesonide nasal aerosol 37 mcg or 74 mcg or placebo for 2 weeks of treatment) and Follow-up. The total duration of subject participation will be approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Gives written informed consent (parent/legal guardian) and assent (from the child), including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Is a male or premenarchal female 6 to 11 years-old at the screening.
* Is in general good health (defined as the absence of any clinically relevant abnormalities as determined by the investigator) based on screening physical examination and medical history.
* Has a history of SAR to any relevant dominant seasonal allergen for a minimum of one to two years immediately preceding the study Screening Visit. The SAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past and is expected to require treatment throughout the entire study period.
* Has a demonstrated sensitivity to a relevant dominant seasonal allergen known to induce SAR based on a documented result with a standard skin prick test either within 12 months prior to screening or performed at the screening visit. A positive test is defined as a wheal diameter at least 3 mm larger than the control wheal (normal saline) for the skin prick test. The subject's positive allergen test must be consistent with the medical history of SAR, and the allergen must be present in the subject's environment throughout the study.
* Subject or parent/guardian must possess an educational level and degree of understanding of English that enables them to communicate suitably with the Investigator and study coordinator as well as accurately complete both the Allergic Rhinitis diary and Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ).

Exclusion Criteria:

* Has a history of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations; recent unhealed nasal biopsy; nasal trauma; or nasal ulcers or perforations. Surgery and atrophic rhinitis or rhinitis medicamentosa are not permitted within the 120 days prior to the screening visit.
* Has evidence of infection, significant anatomic abnormality, ulceration of the mucosa, blood in the nose, or any other clinically relevant finding on nasal examination at the screening visit.
* Has nasal jewelry
* Has participated in any investigational drug trial within the 30 days preceding the screening visit or is planning participation in another investigational drug trial at any time during this trial.
* Has a known hypersensitivity to any corticosteroid or any of the excipients in the formulation of ciclesonide.
* Has a history of a respiratory infection or disorder, including but not limited to bronchitis, pneumonia, influenza, and severe acute respiratory syndrome (SARS), within the 14 days preceding the screening visit.
* Has active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta-agonists and any controller drugs (eg, theophylline, leukotriene antagonists); intermittent use (≤ 3 uses per week) of inhaled short-acting beta-agonists is acceptable. Use of short-acting beta agonists for exercise induced bronchospasm will be allowed.
* Plans to travel outside the study area (the known pollen area for the investigative site) for 2 or more consecutive days between Randomization Visit and the final Treatment Visit.
* Plans to leave the study area (the known pollen area for the investigative site) for longer than 24 hours during the Single-blind Placebo Run-in period.
* Is expecting to use any disallowed concomitant medications during the treatment period.
* Is planning initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the screening visit and use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
* Has nonvaccinated exposure to or active infection with chickenpox or measles within the 21 days preceding the screening visit.
* Initiates pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or plans a dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to screening and use of a stable (maintenance) dose during the study period may be considered for inclusion.
* Is a child or relative of any clinical investigator or site personnel, even those who are not directly involved in this study.
* Has any of the following conditions that are judged by the investigator to be clinically significant and/or to affect the subject's ability to participate in the clinical trial: impaired hepatic function; history of ocular disturbances, eg, glaucoma or posterior subcapsular cataracts or herpes simplex; any systemic infection hematological (including anemia), hepatic, renal, endocrine disease; gastrointestinal disease; malignancy (excluding basal cell carcinoma); current neuropsychological condition with or without drug therapy. Any behavioral condition that could affect subject's ability to accurately report symptoms to the caregiver such as developmental delay, attention deficit disorder, and autism.
* Has any condition that, in the judgment of the investigator, would preclude the subject from completing the protocol with capture of the assessments as written.
* Has received ciclesonide nasal aerosol in a previous clinical trial

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 847 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (66):
- United States (66):
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - San Jose Multispecialty Medical Group, Inc, Baldwin Park, California
  - WCCT Global, LLC, Costa Mesa, California
  - Premier Health Research Center, Downey, California
  - Allergy, Asthma, Brochitis and Immunology Assoc Medical Group, Fountain Valley, California
  - Pediatric Care Medical Group, Inc., Huntington Beach, California
  - Pediatric Care Medical Group, Huntington Beach, California
  - Allergy and Asthma Associates of Southern California, Mission Viejo, California
  - CHOC, PSF, AMC, Division of Allergy, Asthma, and Immunology, Orange, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Capital Allergy & Respiratory Disease Center, Sacramento, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy & Asthma Medical Group and Research Center, APC, San Diego, California
  - Bensch Research Associates, Stockton, California
  - Asthma & Allergy Associates, PC, Colorado Springs, Colorado
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, PC, Denver, Colorado
  - Northeast Georgia Research Center, Gainesville, Georgia
  - DataQuest Medical Research, LLC, Lawerenceville, Georgia
  - Atlanta Allergy & Astma Clinic, Marietta, Georgia
  - Aeroallergy Research Laboratories of Savannah, Inc, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Alzein Pediatrics, Evergreen Park, Illinois
  - Sneeze, Weeze, & Itch Associates, Normal, Illinois
  - Gordon D. Raphael, MD, Berthesda, Maryland
  - Clinical Research Institute, Plymouth, Minnesota
  - Creighton University Medical Center, Omaha, Nebraska
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Catalyst Medical Center, Fargo, North Dakota
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Baker Allergy Asthma and Dermatology Research Center LLC, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - Asthma, Nasal Disease & Allergy Research Center of New England, Providence, Rhode Island
  - National Allergy, Asthma, and Uticaria Centers of Charleston, PA, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - DCT - Anchor, LLC dba Discovery Clinical Trials, Arlington, Texas
  - Discovery Clinical Trials, Arlington, Texas
  - Benchmark Research, Austin, Texas
  - Isis Clinical Research, LLC, Austin, Texas
  - Sirius Clinical Research LLC, Austin, Texas
  - TTS Research Center, Boeme, Texas
  - Research Across America, Carroliton, Texas
  - Dallas Allergy Immunology Research, Dallas, Texas
  - Pharmaceutical Research and Consulting, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Benchmark Research, Fort Worth, Texas
  - Kerrville Research Associates, Kerrville, Texas
  - Live Oak Allergy and Asthma Clinic, Live Oak, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - ACRC Trials, Plano, Texas
  - North Texas Family Medicine, Plano, Texas
  - Benchmark Research, San Angelo, Texas
  - Sun Research Institute, San Antonio, Texas
  - DCT - Barlite Dba Discovery Clinical Trials, San Antonio, Texas
  - Allergy and Asthma Research Center, PA, San Antonio, Texas
  - San Antonio Ear, Nose & Throat Research, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - DCT-Westover Hills, Dba Discovery Clinical Trials, San Antonio, Texas
  - Pediatric Healthcare of Northwest Houston, Tomball, Texas
  - Allergy & Asthma Care of Waco, Waco, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - Ericksen Research and Development, Clinton, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Started | 283 | 282 | 282
Completed | 269 | 269 | 273
Not Completed | 14 | 13 | 9
Not completed — Adverse Event | 3 | 4 | 1
Not completed — Lost to Follow-up | 3 | 2 | 5
Not completed — Protocol Violation | 5 | 5 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg | Total
Number analyzed (Participants) | 283 | 282 | 282 | 847
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 283 | 282 | 282 | 847
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (1.72) | 8.5 (1.64) | 8.7 (1.65) | 8.6 (1.65)
Age, Customized [Number; unit: participants]
  6-8 Years | 131 | 123 | 120 | 374
  9-11 Years | 152 | 159 | 162 | 473
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 123 | 120 | 374
  Male | 152 | 159 | 162 | 473
Region of Enrollment [Number; unit: participants]
  United States | 283 | 282 | 282 | 847

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Subject Reported AM and PM Reflective Total Nasal Symptom Scores (rTNSS) Over the 2-week Double-blind Treatment Period
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent 1 = mild 2 = moderate 3 = severe. Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0 - 2
Population: n = number of ITT subjects in treatmentgroup with completed assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 280 | 279 | 281
units on a scale | -1.63 (0.133) | -1.73 (0.133) | -1.61 (0.133)

2. Secondary Outcome: Change From Baseline in Average Daily Subject-reported AM and PM Instantaneous Total Nasal Symptom Scores (iTNSS) Over the 2-week Double-blind Treatment Period
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent 1 = mild 2 = moderate 3 = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0 - 2
Population: n = number of ITT subjects in treatment group with completed assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 278 | 281 | 280
units on a scale | -1.32 (0.125) | -1.48 (0.125) | -1.35 (0.125)

3. Secondary Outcome: Change From Baseline in Average Daily Subject-reported AM and PM Reflective Total Ocular Symptom Scores (rTOSS) Over the 2-week Double-blind Treatment Period.
Description: TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TOSS symptom scores assess symptoms over the previous 12-hour time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0 - 2
Population: n = number of ITT subjects in treatment group with completed assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 279 | 281 | 279
units on a scale | -0.84 (0.090) | -0.69 (0.090) | -0.79 (0.090)

4. Secondary Outcome: Change From Baseline in the Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) Overall Score at the End of the Double-blind Treatment Period.
Description: PRQLQ was developed to measure the functional problems (physical, emotional, and social) that are most troublesome to children with rhinoconjunctivitis. The PRQLQ has 23 questions in 5 domains (nose symptoms, eye symptoms, practical problems, activity limitation, and other symptoms). Children recalled how they were during the previous week and responded to each question on a 7-point scale (0 = not bothered to 6 = extremely bothered or 0 = none of the time to 6 = all of the time) for a total possible score of 138. The overall PRQLQ score is the mean of all 23 responses and the individual domain scores are the means of the items in those domains.
Time Frame: Weeks 0 - 2
Population: n = number of ITT subjects in treatment group with completed assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 278 | 279 | 279
units on a scale | -0.41 (0.055) | -0.43 (0.055) | -0.51 (0.054)

5. Secondary Outcome: Change From Baseline in Average Daily Subject Reported AM Instantaneous Total Nasal Symptom Scores (iTNSS) Over the 2-week Double-blind Treatment Period
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions assessed in the AM. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent 1 = mild 2 = moderate 3 = severe in the AM. Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0 - 2
Population: n = number of ITT subjects in treatment group with completed assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 278 | 281 | 279
units on a scale | -1.27 (0.126) | -1.48 (0.126) | -1.34 (0.126)

6. Secondary Outcome: Change From Baseline in Average Daily Subject-reported AM and PM Instantaneous Total Ocular Symptom Scores (iTOSS) Over the 2-week Double-blind Treatment Period.
Description: TOSS is the sum of individual ocular symptoms of itching, tearing, and redness. Subjects assess each individual symptoms on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, TOSS ranges from 0-9 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TOSS symptom scores assess symptoms over the previous 10 minute time interval. Difference was calculated as the two week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement
Time Frame: Weeks 0 - 2
Population: n = number of ITT subjects in treatment group with completed assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 279 | 281 | 279
units on a scale | -0.71 (0.088) | -0.57 (0.088) | -0.66 (0.088)

7. Secondary Outcome: Time to Maximal Effect in the AM and PM Reflective Total Nasal Symptom Scores (rTNSS) Over the 2-week Double-blind Treatment Period
Description: The time to maximal effect, defined as the number of days until the first treatment day on which the estimated difference between ciclesonide nasal aerosol and placebo was at least 90% of the largest estimated difference, was based on the analyses of change from baseline in the average of AM and PM rTNSS scores for each day. The time to achieve at least 90% of these estimated differences is presented.
Time Frame: Weeks 0 - 2
Measure: Number; unit: Days
Arm/Group | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 282 | 282
Days | 2 | 13

8. Secondary Outcome: Number of Subjects Experiencing Treatment-emergent AEs
Description: Treatment-Emergent Adverse Events Occurring in ≥ 2% of Subjects in Any Treatment Group (ITT Population)
Time Frame: Weeks 0 - 3
Measure: Number; unit: participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 282
participants
  PYREXIA | 4 | 5 | 7
  HEADACHE | 9 | 14 | 10
  COUGH | 6 | 4 | 4
  EPISTAXIS | 10 | 12 | 6

9. Secondary Outcome: Percentage of Subjects Experiencing Treatment-emergent AEs
Description: Treatment-Emergent Adverse Events Occurring in ≥ 2% of Subjects in Any Treatment Group (ITT Population)
Time Frame: Weeks 0 - 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 282
Percentage of participants
  PYREXIA | 1.4 | 1.8 | 2.5
  HEADACHE | 3.2 | 5.0 | 3.5
  COUGH | 2.1 | 1.4 | 1.4
  EPISTAXIS | 3.5 | 4.3 | 2.1

10. Secondary Outcome: Treatment-emergent AEs Causing Study Medication Discontinuation
Time Frame: Weeks 0 - 3
Measure: Number; unit: participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 282
participants
  Application site pain | 0 | 0 | 1
  Hypersensitivity | 0 | 1 | 0
  Pharyngitis streptococcal | 0 | 1 | 0
  Allergic respiratory symptom | 1 | 0 | 0
  Asthma | 1 | 2 | 0
  Rhinitis seasonal | 1 | 0 | 0

11. Secondary Outcome: Number of Subjects Experiencing Treatment-emergent Nasal AEs, Including Epistaxis, Nasal Ulceration, and Nasal Perforation
Time Frame: Weeks 0 - 3
Measure: Number; unit: participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 282
participants
  Acute sinusits | 0 | 1 | 1
  Application site burn | 1 | 0 | 0
  Application site pain | 3 | 4 | 3
  Epistaxis | 10 | 12 | 6
  Mucosal erosion | 0 | 1 | 0
  Mucosal excoriation | 1 | 0 | 0
  Mucosal haemorrhage | 0 | 1 | 0
  Nasal congestion | 1 | 0 | 0
  Nasal discomfort | 0 | 5 | 0
  Nasal dryness | 0 | 0 | 1
  Nasal mucosal disorder | 1 | 1 | 0
  Nasal septum ulceration | 0 | 0 | 1
  Rhinalgia | 1 | 0 | 0
  Rhinitis seasonal | 1 | 1 | 0
  Scab | 0 | 1 | 0
  Scratch | 1 | 0 | 0
  Sinus headache | 1 | 0 | 0
  Sinus lesion | 1 | 0 | 0
  Sneezing | 0 | 0 | 1

12. Secondary Outcome: Percentage of Subjects Experiencing Treatment-emergent Nasal AEs, Including Epistaxis, Nasal Ulceration, and Nasal Perforation
Time Frame: Weeks 0 - 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 282
Percentage of participants
  Acute sinusits | 0 | 0.4 | 0.4
  Application site burn | 0.4 | 0 | 0
  Application site pain | 1.1 | 1.4 | 1.1
  Epistaxis | 3.5 | 4.3 | 2.1
  Mucosal erosion | 0 | 0.4 | 0
  Mucosal excoriation | 0.4 | 0 | 0
  Mucosal haemorrhage | 0 | 0.4 | 0
  Nasal congestion | 0.4 | 0 | 0
  Nasal discomfort | 0 | 1.8 | 0
  Nasal dryness | 0 | 0 | 0.4
  Nasal mucosal disorder | 0.4 | 0.4 | 0
  Nasal septum ulceration | 0 | 0 | 0.4
  Rhinalgia | 0.4 | 0 | 0
  Rhinitis seasonal | 0.4 | 0.4 | 0
  Scab | 0 | 0.4 | 0
  Scratch | 0.4 | 0 | 0
  Sinus headache | 0.4 | 0 | 0
  Sinus lesion | 0.4 | 0 | 0
  Sneezing | 0 | 0 | 0.4

ADVERSE EVENTS:
Time Frame: Weeks 0 to 3
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Serious Adverse Events (participants affected / at risk) | 0/283 | 1/282 | 0/282
Other Adverse Events (participants affected / at risk) | 25/283 | 31/282 | 24/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=283) | Ciclesonide Nasal Aerosol 37mcg (N=282) | Ciclesonide Nasal Aerosol 74 mcg (N=282)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=283) | Ciclesonide Nasal Aerosol 37mcg (N=282) | Ciclesonide Nasal Aerosol 74 mcg (N=282)
PYREXIA (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 7 (7)
HEADACHE (Nervous system disorders) | 9 (12) | 14 (15) | 10 (10)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 4 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 12 (17) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.